CLINICAL TRIAL: NCT01023997
Title: Central Corneal Thickness in Patients With Exfoliation Syndrome, Exfoliative Glaucoma, Exfoliative Glaucoma, Primary Open-angle Glaucoma and Ocular Hypertension
Brief Title: Central Corneal Thickness in Glaucoma
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, AGP Konstas, Professor in Ophthalmology, Aristotle University Of Thessaloniki
Other Study IDs: A3502
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Exfoliation Syndrome
Keywords: corneal thickness; exfoliation
MeSH Terms: conditions — Exfoliation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- primary open-angle glaucoma
- ocular hypertension patients
- normal controls
- Exfoliation patients: patients with exfoliation syndrome or exfoliative glaucoma

SUMMARY:
The purpose of this study is to compare the central corneal thickness measurement in patients with exfoliation syndrome, exfoliative glaucoma, primary open-angle glaucoma, ocular hypertension and normal controls and to evaluate the value of corneal thickness in the diagnosis and management of glaucoma.

DETAILED DESCRIPTION:
To compare the central corneal thickness measurement in patients with exfoliation, primary open-angle glaucoma, ocular hypertension and normal controls and to evaluate the value of corneal thickness in the diagnosis and management of glaucoma. Prospective study in progress. Randomly selected patients undergo a comprehensive ophthalmic exam which includes 2 separate pachymetry measurements in 2 different examinations at the same time of the day (10:00 am) with 3 different pachymeters. The values obtained are correlated with a number of other glaucoma parameters. A thinner cornea may represent a specific attribute and an additional risk factor for patients with exfoliation. Evaluation of corneal thickness is an important exam in the management of patients with exfoliation.

ELIGIBILITY:
Inclusion Criteria:

* Exfoliation material on pupil
* Intraocular pressure below 21 mm Hg without glaucomatous damage
* Intraocular pressure above 21 mm Hg without glaucomatous damage
* Raised intraocular pressure with glaucomatous damage

Exclusion Criteria:

* Corneal disorders
* History of trauma
* Evidence of corneal abnormality that may influence IOP
* Contact lens use
* Corneal surgery

Ages: 25 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals with and without exfoliation
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2008-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
central corneal thickness | Morning measurement (10:00-11:00)

SECONDARY OUTCOMES:
Visual field, scanning laser polarimetry | 10:00-11:00

CONTACTS AND LOCATIONS:
Overall Officials: Kostantinos Kaltsos, MD, PhD, Study Director — 1st University Dept of Ophthalmology
Locations (1):
- Glaucoma Unit, 1st University Department of Ophthalmology, Thessaloniki, Greece